CLINICAL TRIAL: NCT02310802
Title: A Phase 2, Double-blind, Dose-finding, Placebo-controlled Study to Assess the Safety and Efficacy of a Single Oral Administration of OBE001 to Improve Embryo Implantation Following IVF or ICSI
Brief Title: OBE001 Phase 2 Dose-finding Study Versus Placebo in Women Undergoing Embryo Transfer in the Context of IVF-ICSI
Acronym: IMPLANT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-OBE001-013
Record Dates: First submitted 2014-11-19; First posted 2014-12-08 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Infertility
Keywords: IVF; ICSI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- OBE001 dose 1 (Experimental)
  Interventions: Drug: OBE001 dose 1
- OBE001 dose 2 (Experimental)
  Interventions: Drug: OBE001 dose 2
- OBE001 dose 3 (Experimental)
  Interventions: Drug: OBE001 dose 3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OBE001 dose 1 — OBE001 dispersible tablets for single oral administration
  Arms: OBE001 dose 1
Drug: OBE001 dose 2 — OBE001 dispersible tablets for single oral administration
  Arms: OBE001 dose 2
Drug: OBE001 dose 3 — OBE001 dispersible tablets for single oral administration
  Arms: OBE001 dose 3
Drug: Placebo — Placebo dispersible tablets for single oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the increase in clinical pregnancy rate after administration of a range of single oral doses of OBE001, an oral oxytocin antagonist, compared to placebo.

DETAILED DESCRIPTION:
The study is a prospective, dose-finding, randomised, parallel group, double-blind, placebo-controlled study investigating the efficacy and the safety of the oxytocin receptor antagonist OBE001 in 240 women undergoing embryo transfer following IVF or ICSI.

The four-arm study (OBE001 dose 1, dose 2, dose 3, and placebo) design will allow evaluation of a possible dose-dependent pattern of action of OBE001 and, simultaneously, comparison of active compound with placebo with regard to both efficacy and safety.

ELIGIBILITY:
Key Inclusion Criteria

1. Women with medically indicated IVF or ICSI using her own oocytes.
2. GnRH antagonist protocol, a single injection of hCG for triggering final follicular maturation and luteal phase support with vaginal micronized progesterone.
3. Evidence of uterine contractions by transvaginal ultrasound at baseline.

Key Exclusion Criteria

1. Blastocyst stage or frozen-thaw transfers
2. Clinically significant abnormalities in ECG, vital signs, physical examination or clinical laboratory results
3. Severe endometriosis and/or adenomyosis or risk of ovarian hyper stimulation syndrome

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 247 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
EFFICACY ENDPOINTS Percentage of women with an intra-uterine pregnancy with positive embryo heart-beat | about 6 weeks post ET day
  Percentage of women with an intra-uterine pregnancy with positive embryo heart-beat at about 6 weeks post ET day.

SECONDARY OUTCOMES:
EFFICACY ENDPOINTS Percentage of women with positive blood pregnancy test | 14 days post OPU day
  Percentage of women with positive blood pregnancy test at 14 days post OPU day.
EFFICACY ENDPOINTS Percentage of women with an intra-uterine pregnancy with positive embryo heart-beat | 10 weeks post OPU day
  Percentage of women with an intra-uterine pregnancy with positive embryo heart-beat at 10 weeks post OPU day.
EFFICACY ENDPOINTS The embryo-implantation rate | 6 weeks post ET day
  The embryo-implantation rate defined as the number of intra-uterine embryos with positive heart-beat at 6 weeks post ET day divided by the number of embryos transferred
EFFICACY ENDPOINTS Change from baseline to the time of ET in the rate of uterine contractions | at 3.5 hours after dose administration
  Change from baseline to the time of ET in the rate of uterine contractions (UC/min).

OTHER OUTCOMES:
SAFETY ENDPOINTS Treatment emergent adverse events frequency and severity | up to 10 weeks post OPU day
  Treatment emergent adverse events frequency and severity
SAFETY ENDPOINTS (Haematology and biochemistry assessments) | 14 days post OPU day
  Haematology and biochemistry assessments at screening and at visit V3 (14 days post OPU day)
PHARMACOKINETIC ENDPOINTS Plasma levels of OBE001 | at 3.5 hours after dose administration
  Plasma levels of OBE001
PHARMACOKINETIC-PHARMACODYNAMIC ENDPOINTS :Uterine contractions relationship to OBE001 plasma levels and pregnancy rate | up 10 weeks post OPU day
  Uterine contractions relationship to OBE001 plasma levels and pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Director, Study Director — ObsEva SA
Locations (18):
- Brussels, Belgium
- Czechia (4):
  - Hradev Kralove
  - Olomouc
  - Prague
  - Zlín
- Denmark (2):
  - Copenhagen
  - Hvidovre
- Poland (4):
  - Bialystok
  - Katowice
  - Szczecin
  - Warsaw
- Spain (6):
  - Alicante
  - Barakaldo
  - Barcelona
  - Bilbao
  - Seville
  - Vigo
- London, United Kingdom

REFERENCES:
- [Derived] Griesinger G, Blockeel C, Pierzynski P, Tournaye H, Visnova H, Humberstone A, Terrill P, Pohl O, Garner E, Donnez J, Loumaye E. Effect of the oxytocin receptor antagonist nolasiban on pregnancy rates in women undergoing embryo transfer following IVF: analysis of three randomised clinical trials. Hum Reprod. 2021 Mar 18;36(4):1007-1020. doi: 10.1093/humrep/deaa369. PMID 33534895